CLINICAL TRIAL: NCT07392619
Title: Evaluation of the Effect of Acupressure Applied to Older Adults With Painful Diabetic Peripheral Neuropathy on Neuropathic Symptoms, Balance Confidence, Fear of Falling, and Quality of Life:
Brief Title: The Effect of Acupressure on Symptoms in Elderly Adults With Painful Diabetic Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Nigde Omer Halisdemir Univ.
Record Dates: First submitted 2025-12-11; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Painful Diabetic Peripheral Neuropathy (PDPN); Acupressure
Keywords: diabetic neuropathic symptoms; balance confidence; fear of falling; quality of life; olderly individuals; acupressure
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: This project will be conducted using a mixed methodology integrating quantitative and qualitative methods. Elderly individuals will be randomly assigned to an acupressure or placebo control group. The acupressure group will receive a total of 10 sessions of acupressure over one month.The study will employ a double-blind design. Participants will be randomly assigned to either the acupressure or placebo acupressure groups upon volunteering, with an equal chance of being assigned to either group. A standardized administration procedure/protocol will be used to prevent differences in administration between groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (Active Comparator): The acupressure group will receive a total of 10 sessions of acupressure over one month.
  Interventions: Other: acupressure
- placebo control (Placebo Comparator): For individuals in the placebo (sham) acupressure group, placebo (sham) acupressure will be applied away from the designated acupoint. The number, duration, frequency and application protocol of sessions in the placebo acupressure group will be the same as in the acupressure group.
  Interventions: Other: placebo acupressure

INTERVENTIONS:
Other: acupressure — Acupressure is a method based on the correction of yang and yin imbalances in the body by manipulating points located on meridians close to the skin. The primary goal of acupressure is to restore the flow of Qi (Chi/Chi/Chi), the energy that constantly flows throughout the body. From a practical perspective, acupressure requires no special equipment and is non-invasive compared to other treatment techniques.
  Other Names: placebo acupressure
  Arms: Acupressure
Other: placebo acupressure — Individuals in the placebo (sham) acupressure group will receive placebo (sham) acupressure distant from the designated acupoint.
  Arms: placebo control

SUMMARY:
This project aims to evaluate the effects of acupressure applied to elderly individuals with painful diabetic peripheral neuropathy (DPN) on neuropathic symptoms, balance confidence, fear of falling, and quality of life. This project will be conducted using a mixed methodology integrating quantitative and qualitative methods. Elderly individuals will be randomly assigned to an acupressure or placebo control group. The acupressure group will receive a total of 10 sessions of acupressure over one month. Outcome measures include assessments of neuropathic pain and symptoms, balance confidence, fear of falling, and quality of life. Appropriate statistical tests will be used to analyze the quantitative data obtained from the study, while content analysis will be used for the qualitative data.

DETAILED DESCRIPTION:
To avoid ignoring the increasing disease burden, decreased productivity, and other problems of elderly individuals, it is important to carefully consider GETAT (Traditional and Complementary Medicine) approaches that may be beneficial in controlling their multiple symptoms in this specific group.

This study aims to evaluate the effect of acupressure on neuropathic symptoms, balance confidence, fear of falls, and quality of life in elderly individuals with Painful Diabetic Peripheral Neuropathy (PDN).

This research will be conducted at Niğde Training and Research Hospital. The research population consists of individuals who participate in planned visits to the Internal Medicine outpatient clinics of Niğde Training and Research Hospital, have a prior diagnosis of DM, and have been diagnosed with DPN by a specialist physician.

Individuals in the acupressure group will participate in a program consisting of a total of 10 sessions over one month. Each session will consist of preparation, application, and termination steps.

The acupuncture points to be applied in this research were determined by an experienced acupuncture specialist and the researcher, according to GETAT methods and in line with the literature.

The number, duration, frequency, and application protocol of sessions in the placebo-acupressure group will be the same as in the acupressure group. The only difference between the two groups is the location of the points.

The study will be conducted in accordance with the 1964 Helsinki Declaration. Research will commence after the purpose and methodology of the study are explained to the participants, anonymity and confidentiality are guaranteed, their willingness to participate is confirmed, and participants provide their BOGs (Brain Stability Questionnaire).

Outcome measures include assessment of neuropathic pain and symptoms, balance confidence, fear of falling, and quality of life. Appropriate statistical tests will be used to analyze quantitative data, and content analysis will be used for qualitative data.

ELIGIBILITY:
Inclusion Criteria:

Elderly individuals aged 65 years and older

No sensory impairment that would hinder communication

Cognitively capable of answering questions

Able to walk independently or with an assistive device

Have not previously received acupressure therapy for DPN

Diagnosed with diabetic peripheral neuropathy (DPN) by a physician

No orthopedic problems

Provide informed consent

Exclusion Criteria:

Not providing informed consent

History of non-diabetic neuropathy

Physician-diagnosed advanced cardiovascular, kidney, or liver disease

Bleeding tendency

Cerebrovascular disease

History of medical conditions such as retinopathy or nephropathy

Presence of open wounds, ulcers, or orthopedic problems on the feet

Inability to walk independently

Not voluntarily agreeing to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-12-30 (Estimated); Primary Completion 2027-09-05 (Estimated); Study Completion 2028-09-05 (Estimated)

PRIMARY OUTCOMES:
DIABETIC NEUROPATHY SYMPTOM SCORE | 0-4 weeks
  Diabetic neuropathy symptoms will be assessed using the Diabetic Neuropathy Symptom Score (DNS) and reported as a total score (points).The Diabetic Neuropathy Symptom Score will be used to assess participants' diabetic neuropathy symptoms. It consists of four questions related to gait imbalance, neuropathic pain, paresthesia, and numbness. Each question is scored from 0 (none) to 1 (yes), and a total score is calculated. The maximum score is 4 points, and a score of 1 or higher is defined as positive for DPN.
Neuropathic Pain Scale | 0-4 weeks
  Neuropathic pain level will be measured using the Self-Administered Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) questionnaire and reported as a score (points). In this study, the Self-Administered-Leeds Assessment of Neuropathic Symptoms and Signs Pain Score (S-LANSS) will be used to evaluate neuropathic pain. Participants will respond "yes" if the pain symptom is consistent with the description, and "no" if the pain symptom is inconsistent. The total score is scored between 0 and 24. The cutoff value is 12, and if the total score is ≥12, neuropathic mechanisms may be responsible for the pain experienced by the patient.

SECONDARY OUTCOMES:
BALANCE CONFIDENCE SCALE | 0-4 weeks
  Balance confidence in elderly participants will be evaluated using the Activities-specific Balance Confidence (ABC) Scale and reported as a total score (points).One of the tools frequently used to assess fear of falling is the 16-item Activity-Specific Balance Confidence Scale. It is rated from 0 (unsafe) to 100 (completely confident), with a score ranging from 0 to 1600. The total score is divided by 16 to determine the scale score. Higher scores indicate increased balance confidence. A score of <50 out of 100 indicates low physical function, 50-80 indicates moderate physical function, and 80 or above indicates high physical function.
European General Quality of Life Scale (EQ-5D). | 0-4 weeks
  Quality of life will be measured using the EuroQol 5-Dimension (EQ-5D) questionnaire and reported as a total score (points).Individuals' quality of life will be assessed using the European General Quality of Life Scale (EQ-5D). This is a reporting tool that uses six questions to assess individuals' overall quality of life, independent of their current medical condition. The scale has five dimensions, and each dimension has five levels. The EQ-5D descriptive system measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels corresponding to "no problem", "mild problem", "moderate problem", "severe problem", and "extreme problem". In the EQ-VAS, quality of life scores range from 0 to 100, with 0 representing the worst health condition and 100 representing the best health condition. As the scale score increases, the perception of health increases positively.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan TAŞCI, Prof. Dr., Study Director — TC Erciyes University

IPD SHARING:
Plan to Share IPD: No
To protect personal data, individual participant data will not be shared. However, study results will be published as an article based on the individuals' voluntary consent.